CLINICAL TRIAL: NCT05809414
Title: Amantadine and Transcranial Magnetic Stimulation for Treating Fatigue in Multiple Sclerosis: Phase III Study, Controlled, Randomized, Crossed Over and Double Blind.
Brief Title: Amantadine and Transcranial Magnetic Stimulation for Treating Fatigue in Multiple Sclerosis
Acronym: FETEM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Jorge Matías-Guiu, Principal Investigator, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: FETEM
Record Dates: First submitted 2023-03-20; First posted 2023-04-12 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Multiple Sclerosis; Fatigue
Keywords: Amantadine; Multiple Sclerosis; Fatigue; Transcranial Magnetic Stimulation (TMS); Modified Fatigue Impact Scale (MFIS)
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Transcranial Magnetic Stimulation; Amantadine; Magnesium

STUDY DESIGN:
Intervention Model Description: All patients will receive all possible combinations (TMS+placebo, TMS+amantadine, TMS sham+amantadine, TMS sham+placebo), the only difference being the sequence in which they are administered.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Amantadine (Experimental)
  Interventions: Drug: Amantadine Hydrochloride 100 mg (milligrams) Oral Capsule
- Placebo (Placebo Comparator)
  Interventions: Drug: Amantadine Hydrochloride 100 mg (milligrams) Oral Capsule
- TMS (Experimental)
  Interventions: Device: Transcranial Magnetic Stimulation
- TMS sham (Sham Comparator)
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — TMS is a technique for electrical stimulation of brain tissue by generating a magnetic field, which modulates neural activity at the stimulation site and in interconnected neural networks.
  The treatment will be applied to the left dorsolateral prefrontal region. Each patient will receive 3 sessions per week of approximately 10 minutes for 6 weeks.
  In the case of TMS sham, a placebo coil will be used, which is indistinguishable from the therapeutic one. In addition, the sessions will be carried out with the same frequency, so the patient will be unaware of the treatment they are receiving.
  Other Names: TMS
  Arms: TMS; TMS sham
Drug: Amantadine Hydrochloride 100 mg (milligrams) Oral Capsule — It will be used at a dose of 100 mg, 1 capsule a day for 1 week, followed by 2 daily doses of 100 mg until completing 6 weeks in total. After completing the treatment phase, the dose will be de-escalated (1 capsule a day for 5 days and discontinued).
  In the case of placebo amantadine capsules, they will have the same organoleptic characteristics as amantadine. The start, maintenance and de-escalation pattern will be identical.
  Arms: Amantadine; Placebo

SUMMARY:
Multiple Sclerosis (MS) is the most frequent cause of non-traumatic disability in people under 55 years of age. Fatigue is the most frequent and disabling symptom in the disease, and for which there is no effective treatment. Among the proposed drugs, amantadine is the one that could be most useful, although up to now it has not been adequately demonstrated due to a lack of sufficiently powerful and methodologically appropriate clinical trials. Transcranial magnetic stimulation (TMS) has recently been proposed as a useful treatment for fatigue in MS in preliminary studies.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is the most frequent cause of non-traumatic disability in people under 55 years of age. Fatigue is the most frequent and disabling symptom in the disease, and for which there is no effective treatment. Among the proposed drugs, amantadine is the one that could be most useful, although up to now it has not been adequately demonstrated due to a lack of sufficiently powerful and methodologically appropriate clinical trials. Transcranial magnetic stimulation (TMS) has recently been proposed as a useful treatment for fatigue in MS in preliminary studies.

The main objective of the study is to evaluate the change in the severity of fatigue in MS patients undergoing treatment with amantadine, TMS and both in combination, compared to placebo. A randomized, placebo-controlled, crossover, double-blind clinical trial will be conducted. As secondary objectives, changes in cognition, depression and quality of life will be evaluated. For all this, the reference scales adequately validated for each of the objectives will be used.

ELIGIBILITY:
Inclusion Criteria:

1. Expanded Disability Status Scale mark 1.5 - 4.5
2. Fatigue Severity Scale > 4
3. Beck Depression Inventory < 30
4. No relapse for, at least, three month prior to screening
5. Drug washout period = 4 weeks for any fatigue aimed drug
6. Patient capable to sign the informed consent

Exclusion Criteria:

1. Fatigue causing disease other than multiple sclerosis:

   1. sleep apnea
   2. other autoimmune disease that could be explain the fatigue.
   3. endocrine autoimmune disease if the blood test is not in range in the last 6 month.
   4. patient with diagnosis of chronic fatigue
   5. Patient with high blood pressure out of range or decompensated heart failure or New York Heart Association (NYHA) 3-4.
2. Secondary Epilepsy or neuropathic chronic pain which requires continuous treatment.
3. Contraindication for trial treatment:

   1. Some kind of magnetic metal.
   2. Epilepsy antecedents.
   3. Any drugs that could decrease the seizure threshold
   4. Amantadine sensitivity
   5. Cardiopathy disease, severe kidney failure, Angle-closure glaucoma
4. Breastfeeding, pregnancy, or pregnancy planning phase in the next year. Of childbearing potential and willing to use an acceptable method of contraception during the study period.
5. Patient with a terminal disease with no more than one year life expectancy.
6. Patient has been treated for a maligned disease in the past three years.
7. A scheduled surgery in the course of the trials.
8. Any condition that a member of research team consider could affect to participation/follow up patient.
9. Alcoholic o toxics condition in the last year.
10. Major mental disorders
11. Poor communication skills or poor cognitive condition.
12. Other trial participation in the previous 4 month.
13. Use a chronic drug that could interfere in the clinical outcome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
To assess the fatigue severity | 6 weeks after starting treatment
  To compare the effect of TMS and amantadine alone or in combination therapy compared with placebo on fatigue determined using the Modified Fatigue Impact Scale (Total MFIS score: Range from 0 to 84, from minimal to severe fatigue).

SECONDARY OUTCOMES:
To assess the cognitive condition | 6 weeks after starting treatment
  To compare the effect of TMS and amantadine alone or in combination therapy compared to placebo on cognition determined by the Symbol Digit Modalities Test (SDMT).
To assess the depression condition | 6 weeks after starting treatment
  To compare the effect of TMS and amantadine alone or in combination therapy compared to placebo on depression measured using the Beck Depression Inventory Scale (BDI-II score: Range from 0 to 63, from minimal to severe depression).
To assess the quality of life | 6 weeks after starting treatment
  To compare the effect of TMS and amantadine alone or in combination therapy compared to placebo on the quality of life determined by the Short Form 12 Mental Health scale (SF-12 score: Range from 0 to 100, from worse to better physical and mental health functioning).
Safety assessment | 6 months after randomization
  Analyze the incidence of the adverse events detected in each of the branches, whether or not with multiple sclerosis
Cost-effectivity assessment | 6 weeks after starting treatment
  Determine the cost-effectiveness of the different interventions. The total costs of hospitalization and treatment, as well as other health care, will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Matias-Guiu Guia, MD PhD, Principal Investigator — Hospital San Carlos, Madrid
Locations (4):
- Spain (4):
  - Hospital Puerta del Mar, Cadiz
  - Hospital General Gregorio Marañon, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospitalario Universitario Nuestra Señora de la Candelaria, Santa Cruz de Tenerife

IPD SHARING:
Plan to Share IPD: Yes
The data used will be deposited in a suitable repository that will be complied with the requirements of ISCIII and any other applicable national regulations. Due to the data collected retain their personal character and they can be traced back, they will be safeguarded maintaining their integrity and confidentiality. These data cannot be openly shared after the project's completion. The licenses and access permissions will be determined based on the following criteria before the project's completion: a) The guidelines or recommendations of ISCIII. b) The policies established by the data repository to which the data will be sent. c) Possible restrictions on data publication that may arise from applicable protection schemes for the project's results. In any case, the requirements set forth by ISCIII in the funding call received will be complied with, as well as those considered in other applicable regulations. The dataset used will be stored in a locked condition for a period of 5 years.

REFERENCES:
- [Derived] Matias-Guiu JA, Gonzalez-Rosa J, Hernandez MA, Martinez-Gines ML, Portoles A, Perez-Macias N, Benito-Leon J, Padron I, Prieto J, Matias-Guiu J. Amantadine and/or transcranial magnetic stimulation for fatigue associated with multiple sclerosis (FETEM): study protocol for a phase 3 randomised, double-blind, cross-over, controlled clinical trial. BMJ Open. 2024 Jan 4;14(1):e078661. doi: 10.1136/bmjopen-2023-078661. PMID 38176857